CLINICAL TRIAL: NCT00789204
Title: Effectiveness of a "Global Posture Reeducation" Program for Patients With Low Back Pain
Brief Title: Postural Re-education in Low Back Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Paolo Pillastrini, University of Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FB001022008
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2009-09-22 (Estimated); Status verified 2009-09

CONDITIONS: Low Back Pain
Keywords: exercise; low back pain; posture; rehabilitation
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- GPR (Experimental): Global Postural Re-Education
  Interventions: Other: Global Postural Re-education
- SEP (Active Comparator): Standard Exercise Programm
  Interventions: Other: Standard Exercise Training

INTERVENTIONS:
Other: Global Postural Re-education — The treatment in Global Postural Re-education is a global approach that seeks to identify the biomechanical cause of the problem also in other parts of the body and involves actively the patient in the postural change. Using principles like causality, globality and individuality, the treatment consists of the use for one hour of progressive active stretching posture for specific muscular chain that are shortened. Every posture is maintained for 20 minutes with controlled breathing and the use of manual traction
  Other Names: GPR
  Arms: GPR
Other: Standard Exercise Training — The exercise programme included passive lumbar flexion, pelvic tilt, strengthening of flexor muscles, strengthening of extensor muscles, spine mobilization and stretching exercises.
  Other Names: SEP
  Arms: SEP

SUMMARY:
The Global Postural Re-Education is a global approach for the treatment of musculoskeletal disease. Using specific progressive posture for stretching particular shortened chain muscle the method wants to equilibrate the never-ending war between static and dynamic muscles by guiding the patient in a particular breathing pattern to maintain a correct posture and feeling it.

DETAILED DESCRIPTION:
In some countries there is a physical therapy method called "Global Posture Reeducation" (GPR), which was developed by Philippe Emmanuel Souchard based on 20 years of clinical experience.The method consist to balance the miofascial tension probably responsible for an articular overloading. The method stretches the shortened antigravity muscles that are inside a different static muscles chains. GPR is a global approach that search the biomechanics cause in the near areas, and involves actively the patient in the postural and gestural changes.

ELIGIBILITY:
Inclusion Criteria:

* Lumbalgia Diagnosis
* Age 18-80

Exclusion Criteria:

* Migrated hernia
* Calcified disc hernia
* Spondylolisthesis
* Other physiotherapeutic interventions within 6 months of the baseline assessment.
* Surgical operation within six months of baseline
* Cancer syndrome, Neurological and rheumatic diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Roland & Morris Disability Questionnaire | Baseline, 3 months, 6 months

SECONDARY OUTCOMES:
Oswestry Disability Index | Baseline, 3 months, 6 months
Pain Drawing and Visual Analogue Scale (V.A.S.) | Baseline, 3 mounths, 6 months
Fingertip-to-floor test | Baseline, 3 mounths, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Bonetti, Laurea, Principal Investigator
Locations (1):
- Ecm Eur Centro Medico, Rome, Lazio, Italy

REFERENCES:
- [Background] Vanti C, Generali A, Ferrari S, Nava T, Tosarelli D, Pillastrini P. [ General postural rehabilitation in musculoskeletal diseases: scientific evidence and clinical indications]. Reumatismo. 2007 Jul-Sep;59(3):192-201. Italian. PMID 17898878
- [Background] Fernandez-de-Las-Penas C, Alonso-Blanco C, Morales-Cabezas M, Miangolarra-Page JC. Two exercise interventions for the management of patients with ankylosing spondylitis: a randomized controlled trial. Am J Phys Med Rehabil. 2005 Jun;84(6):407-19. doi: 10.1097/01.phm.0000163862.89217.fe. PMID 15905654
- [Background] Hayden JA, van Tulder MW, Malmivaara A, Koes BW. Exercise therapy for treatment of non-specific low back pain. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD000335. doi: 10.1002/14651858.CD000335.pub2. PMID 16034851
- [Derived] Bonetti F, Curti S, Mattioli S, Mugnai R, Vanti C, Violante FS, Pillastrini P. Effectiveness of a 'Global Postural Reeducation' program for persistent low back pain: a non-randomized controlled trial. BMC Musculoskelet Disord. 2010 Dec 16;11:285. doi: 10.1186/1471-2474-11-285. PMID 21162726